CLINICAL TRIAL: NCT04607837
Title: A Randomized, Double Blind, Placebo Controlled, 52 Week Study to Assess the Efficacy and Safety of Etrasimod in Subjects With Moderately Active Ulcerative Colitis
Brief Title: Etrasimod Versus Placebo for the Treatment of Moderately Active Ulcerative Colitis
Acronym: GLADIATOR UC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD334-210; 2020-003507-34 (EudraCT Number); C5041011 (Other: Alias Study Number)
Expanded Access: NCT06025227 (Available)
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Etrasimod; APD334; UC
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod — Etrasimod 2 mg tablet by mouth, once daily up to 52 weeks of treatment
  Other Names: APD334
  Arms: Etrasimod 2 mg
Drug: Placebo — Etrasimod matching placebo tablet by mouth, once daily up to 52 weeks of treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether oral etrasimod is a safe and effective treatment for moderately active ulcerative colitis in adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Ulcerative Colitis (UC) ≥ 3 months prior to screening
* Active UC confirmed by endoscopy
* Moderately active UC defined as a modified Mayo score of 4 to 6 and an endoscopic score ≥ 2 and rectal bleeding score ≥ 1
* Received a surveillance colonoscopy within 12 months before baseline

Exclusion Criteria:

* Severe extensive colitis
* Diagnosis of Crohn's disease or indeterminate colitis or the presence or history of a fistula consistent with Crohn's disease
* Diagnosis of microscopic colitis, ischemic colitis, or infectious colitis
* Hospitalization for exacerbation of UC requiring intravenous steroids within 12 weeks prior to or after screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (285):
- United States (131):
  - Center for Digestive Health (Colonoscopy Location), Dothan, Alabama
  - Digestive Health Specialists, Dothan, Alabama
  - Dothan Eyecare-Dr. Brent McKinley (OCT Location), Dothan, Alabama
  - Pulmonary Associates (Secondary PFT Location), Dothan, Alabama
  - Flowers Hospital (PFT Location), Dothan, Alabama
  - Arizona Retina Institute/ Phoenix Retina Associates(OCT), Peoria, Arizona
  - SimonMed Imaging (Imaging), Peoria, Arizona
  - Sun City Endoscopy (Endoscopy), Sun City, Arizona
  - Euclid Endoscopy Center-El Cajon (Endoscopy procedure only), El Cajon, California
  - Center for Clinical Research (CCR), Irvine, California
  - UCI Gavin Herbert Eye Institute, Irvine, California
  - UCI Gottschalk Medical Plaza, Irvine, California
  - Dr. Raed Al-Naser -Sharp Grossmont outpatient (DLCO procedure only), La Mesa, California
  - Dr. Sally s. Lee in La Mesa (Ophthalmologist procedure only), La Mesa, California
  - Advanced Endoscopy and Pain Center (Colonoscopy), Lancaster, California
  - Advanced Imaging Center (Chest X-Ray), Lancaster, California
  - Antelope Valley Eye Care (Ophthalmologist), Lancaster, California
  - AV Pediatrics, Allergy and Family Medicine (PFT, Physical Exam, ECG Review, Lab Review), Lancaster, California
  - Jatinder S. Pruthi, MD FACG CPI (Physical Exam, ECG Review, Lab Review), Lancaster, California
  - OM Research LLC, Lancaster, California
  - Abraham M. lshaaya MD (X-Ray), Los Angeles, California
  - Entertainment Medical Group, Inc (Main Site, Subject Visits, IP Delivery/Storage, Regulatory,, Los Angeles, California
  - Advanced Vision Care (OCT), Los Angeles, California
  - Century City Endoscopy (Colonoscopy - Nicholas Karyotakis M.D. Endoscopist), Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials, LLC, Los Angeles, California
  - United Surgery Center Murrieta [Endoscopy Only], Murrieta, California
  - United Medical Doctors, Murrieta, California
  - CCR-ICTS Center for Innovative Patient Care, Orange, California
  - UCI Health Eye Care Services (Ophthalmoscopy and OCTs), Orange, California
  - UCI Health H. H. Chao Comprehensive Digestive Disease Center, Orange, California
  - UCI Investigational Drug Services (IDSP - Pharmacy), Orange, California
  - UCI Irvine Medical Center - Pulmonology Services - PFTs, Orange, California
  - ACRC Studies, San Diego, California
  - California Eye Professionals [OCT Only], Temecula, California
  - United Surgery Center Temecula [Endoscopy Only], Temecula, California
  - Front Range Endoscopy Center, Colorado Springs, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Colorado Springs Pulmonary Consultants, PC, Colorado Springs, Colorado
  - The Wright Eye Center (OCT Facility), Colorado Springs, Colorado
  - Colorado Springs Imaging, Colorado Springs, Colorado
  - Florida Advanced Gastroenterology Center - Rahman Nakshabendi MD and Imad Nakshabendi, MD, Brandon, Florida
  - Bay Area Chest Physicians, P.A.,-(Pulmonary Function Test), Clearwater, Florida
  - GASTRO FLORIDA (ADMINISTRATIVE DUTIES etc. CRA visits), Clearwater, Florida
  - West Coast Endoscopy (Colonoscopy Procedures), Clearwater, Florida
  - West Coast Endoscopy Center (Endoscopy Procedures), Clearwater, Florida
  - West Coast Radiology (Chest X-ray), Clearwater, Florida
  - Northwood Vision- Optical Coherence Tomography (OCT), Clearwater, Florida
  - Beraja Medical Institute (OCT), Coral Gables, Florida
  - Juan Barrio, MD (PFT when needed), Coral Gables, Florida
  - The Endoscopy Center (Endoscopy Procedure), Miami, Florida
  - Research Associates of South Florida, Miami, Florida
  - Kendall Endoscopy and Surgery Center (Endoscopy), Miami, Florida
  - Clarin Eye Care Center (OCT/Ophthalmoscopy), Miami, Florida
  - NSB Research, New Smyrna Beach, Florida
  - IMIC Inc, Palmetto Bay, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Larkin Community Hospital (Endoscopy Procedure), South Miami, Florida
  - Absolute Surgical Specialists - Craig Amshel, MD, Sun City Center, Florida
  - SimonMed Imaging, Tampa, Florida
  - Perez Eye Center(OCT & Ophthalmoscopy only), Tampa, Florida
  - Tampa Bay Endoscopy Center(Proctosigmoidoscopy & colonoscopy ONLY), Tampa, Florida
  - Tampa Bay Endoscopy Center, Tampa, Florida
  - Lyracore Health Alliance, Tampa Bay Pulmonology (PFT only), Tampa, Florida
  - Pulmonary and Sleep of Tampa Bay(PFT with DLCO only), Tampa, Florida
  - GCP Clinical Research,LLC, Tampa, Florida
  - LoCicero Medical Group (PFT Procedure Only), Tampa, Florida
  - NewsomEye (OCT only), Tampa, Florida
  - South Tampa Surgery Center, Tampa, Florida
  - GI Alliance (Patients Seen; IP Delivered), Gurnee, Illinois
  - Medical Eye Services LTD (Ophthalmoscopy with OCT), Gurnee, Illinois
  - North Shore Endoscopy Center (Endoscopy), Lake Bluff, Illinois
  - Libertyville Imaging Center (Diagnostic Imaging), Libertyville, Illinois
  - Chevy Chase Endoscopy Center (Endoscopy Facility Only), Chevy Chase, Maryland
  - Chevy Chase Pulmonary Associate (PFT Only), Chevy Chase, Maryland
  - Retina Group of Washington (Ophthalmoscopy and OCT Only), Chevy Chase, Maryland
  - Charter Radiology, Columbia, Maryland
  - Cascades Endoscopy Center, Columbia, Maryland
  - Gastro Center of Maryland, LLC, Columbia, Maryland
  - Kaylani Eye Care ( Optical Coherence Tomography and Opthalmoscopy only), Hanover, Maryland
  - Lung Center (Pulmonary Function Test only), Laurel, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Advantage Diagnostics(X-Ray only), Beachwood, Ohio
  - Geauga Sleep Center(PFT only), Chardon, Ohio
  - UC Health Physicians Office, Cincinnati, Ohio
  - UC Health (Pulmonary Function Testing), Cincinnati, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - The Endoscopy Center of Lake County, Mentor, Ohio
  - Vitreo Retinal Consultants(OCT only), Painesville, Ohio
  - Lake Pulmonary Associates (PFT only), Willoughby, Ohio
  - Retina Specialists of Ohio(OCT only), Willoughby Hills, Ohio
  - West Shore Endoscopy Center, Camp Hill, Pennsylvania
  - Pulmonary and Critical Care Medicine Associates (PFT only), Harrisburg, Pennsylvania
  - Medical Arts Allergy,PC (PFT Only), Harrisburg, Pennsylvania
  - Farrel Opthalmology(OCT only), Harrisburg, Pennsylvania
  - Pinnacle Health Imaging at Tristan (X-Ray only), Harrisburg, Pennsylvania
  - Susquehanna Research Group, Harrisburg, Pennsylvania
  - Harrisburg Eye Associates (OCT only), Harrisburg, Pennsylvania
  - Pulmonary and Critical Care Medicine Associates (PFT only), Lemoyne, Pennsylvania
  - Advanced Radiology Associates (x-Ray only), Edinburg, Texas
  - Texas Retina Associates (OCT Location), Grapevine, Texas
  - Alkek Eye Center Jamail Specialtu Care Center (OCT), Houston, Texas
  - Baylor College of Medicine- Baylor Medical Center, Houston, Texas
  - Baylor College of Medicine-Baylor Medical Center (Chest X-ray location), Houston, Texas
  - Baylor College of Medicine-Baylor Medical Center (IP Storage), Houston, Texas
  - Baylor College of Medicine-Baylor Medical Center (Patients seen address, ECG location, PFT), Houston, Texas
  - Baylor St. Luke's Medical Center Endoscopy- Mc Nair Campus (Endoscopy Location), Houston, Texas
  - Lonestar Endoscopy, Keller, Texas
  - Buena Vista Optical ( OCT only), McAllen, Texas
  - Endoscopy Center at Med Point (Endoscopy only), McAllen, Texas
  - Valley Pulmonary Group (PFT only), McAllen, Texas
  - Envision Imaging, Southlake, Texas
  - Lonestar Endoscopy, Southlake, Texas
  - Texas Digestive Disease Consultants, PLLC d/b/a GI Alliance, Southlake, Texas
  - Christus Trinity Mother Frances Endoscopy Center, Tyler, Texas
  - Christus Trinity Mother Frances Endosopy Center ( endoscopies only), Tyler, Texas
  - Heaton Eye Associates (OCT only), Tyler, Texas
  - Tyler Open MRI (chest x-ray only), Tyler, Texas
  - UT Health East Texas Physicians (pulmonary functions only), Tyler, Texas
  - Citizen Healthplex (PFT), Victoria, Texas
  - Gastro Health & Nutrition - Victoria, Victoria, Texas
  - Surgery Center (Endoscopy), Victoria, Texas
  - Victoria Eye Center (OCT and Opthalmoscopy), Victoria, Texas
  - Harman Eye Center (OCT only), Forest, Virginia
  - Lynchburg Pulmonary Associates, Inc. (PFT only), Lynchburg, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Radiology Consultants of Lynchburg (X-ray only), Lynchburg, Virginia
  - Pacific Northwest Retina, Seattle, Washington
  - Richard Bensinger, MD, Seattle, Washington
  - Swedish Medical Center Investigational Drug Services Pharmacy, Seattle, Washington
  - Swedish Medical Center First Hill Endoscopy Center, Seattle, Washington
  - Swedish Medical Center First Hill, Seattle, Washington
- Australia (12):
  - Queensland Respiratory Services ,Pulse Oceanside Medical{PFT Facility ), Birtinya, Queensland
  - Sunshine Coast Radiology, Birtinya, Queensland
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Buderim Eye Centre( OCT and Ophthalmoscopy Facility), Buderim, Queensland
  - Coral Sea Clinical Research Institute Pty.Ltd, Mackay, Queensland
  - Coastal Digestive Helath Pty. Ltd, Maroochydore, Queensland
  - Dr.Shiran DeSilva Respiratory Clinic (PFT), North Mackay, Queensland
  - Mater Misericordiae Hospital ( Endoscopy), North Mackay, Queensland
  - Queensland X-Ray, North Mackay, Queensland
  - Vision Eye Institute Mackay (OCT), North Mackay, Queensland
  - Austin Health, Heidelberg, Victoria
  - Melbourne Health, Parkville, Victoria
- Belarus (6):
  - Foreign Medical and Pharmaceutical Unitary Enterprise "Medical center "Novoe Zrenie", Grodno
  - Health Care Institution "Grodno City Clinical Hospital #4", Grodno
  - Institution "Gomel Regional Specialized Clinical Hospital", Homyel
  - Institution "Gomel Regional Clinical Hospital", Homyel
  - Health Care Institution "Vitebsk Regional Clinical Specialized Center", Vitebsk
  - Vitebsk Regional Clinical Specialized Center, Vitebsk
- AZ Delta, Roeselare, Belgium
- Bulgaria (13):
  - UMHAT ,,Kanev" AD, Rousse
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - Acibadem City Clinic University Hospital EOOD, Sofia
  - DCC Alexandrovska, EOOD, Sofia
  - UMHAT "Aleksandrovska" EAD (Colonoscopy/Sigmoidoscopy Facility), Sofia
  - UMHAT Aleksandrovska EAD (X-Ray Facility), Sofia
  - UMHAT "Tsaritsa Yoanna-ISUL" EAD, Sofia
  - UMHAT ''Tsaritsa Yoanna-lSUL" EAD (Colonoscopy/ Sigmoidoscopy Facility), Sofia
  - UMHAT Tsaritsa Yoanna - ISUL EAD (X-ray), Sofia
  - University multiprofile hospital for active treatment and emergency medicine N.l Pirogov EAD, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - Acibadem City Clinic University Hospital Eood, Sofia
  - Medical Centre MEDICA Plus OOD, Veliko Tarnovo
- Czechia (14):
  - Gastroenterologicka ambulance, Boskovice
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - VISUS, spol s.r.o., Hradec Králové
  - Gastroenterologicka ordinace MUDr. Pavla Skalova s.r.o., MUDr. Frantisek Sincl s.r.o., Olomouc
  - MUDr. Pavlina Kazinotova, s.r.o., Olomouc
  - PreventaMed s.r.o., Olomouc
  - Gastroenterologie-interna, SPEA, Olomouc
  - Vojenska nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Privatni gastroenterologicka ambulance s.r.o. MUDr. Zdenek Vlk, Prostějov
  - Gastroenterologicka ambulance MUDr. Marcela Vyslouzilova, Přerov
  - Nemocnice Slany, Slaný
  - Poliklinika Slany, spol. s.r.o., Slaný
  - Gatronell s.r.o, Vsetín
- France (3):
  - Centre Hospitalier Universitaire de Genoble Alpes - CHU Michallon, Grenoble
  - Centre Hospitalier Universitaire de Nantes - Hotel-Dieu, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital de l'Archet 2, Nice
- Georgia (10):
  - LLC Academic Pridon Todua Medical Center - LLC Research Institute of Clinical Medicine, Tbilisi
  - LLC Todua Clinic, Tbilisi
  - LTD Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - LTD Vivamedi, Tbilisi
  - LTD Institute of Clinical Cardiology, Tbilisi
  - Medical Center CITO LTD, Tbilisi
  - JSC Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Academician Nikoloz Kipshidze Central University Clinic, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, Tbilisi
- Germany (7):
  - Praxiskooperation Bonn-Euskirchen-Rheinbach-Wesseling, Bonn
  - Florence-Nightingale-Krankenhaus, Düsseldorf
  - OCT: nordBLICK Augenklinik Bellevue, Kiel
  - Universitatsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - OCT: Dr. med. Christopher Kallen, Krefeld
  - OCT: Augenpraxisklinik REMSCHEID, Remscheid
  - Magen-Darm-Zentrum Remscheid, Remscheid
- Hungary (12):
  - Bugat Pal Korhaz, Gyöngyös, Heves County
  - DLCO and ophthalmology tests: Szent Borbala Korhaz, Tatabánya, Komárom-Esztergom
  - Clinfan Szolgaltato Kft., Szekszárd, Tolna County
  - Ophthalmology tests: Tolna Megyei Balassa Janos Korhaz, Szekszárd, Tolna County
  - Ophthalmology tests: Tosho Kft., Budapest
  - Mediszem Kft., Budapest
  - Pulmonary function test: Vasutegeszsegugyi Nonprofit Kozhasznu Kft., Budapest
  - Vasutegeszsegugyi Nonprofit Kozhasznu Kft., Budapest
  - Honvedkorhaz II. telephely, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont (Ophthalmology Tests), Budapest
  - Semmelweis Egyetem Belgyógyászati és Hematológiai Klinika, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
- Israel (4):
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
- Italy (4):
  - Azienda Ospedaliera Saverio De Bellis, Puglia, BARI
  - IRCCS Ospedale San Raffaele, Unita di Gastroenterologia, Milan, Milan
  - Fondazione Policlinico Agostino Gemelli IRCCS, Roma, ROME
  - Ospedale San Bortolo di Vicenza, Gastroenterologia, Vicenza, Veneto
- Poland (20):
  - NSZOZ Termedica - Centrum Badan Klinicznych, Poznan, Greater Poland Voivodeship
  - Allmedica Badania Kliniczne Sp. z o.o. Sp. k., Nowy Targ, Lesser Poland Voivodeship
  - Medicome Sp. z o.o., Oświęcim, Lesser Poland Voivodeship
  - Centrum Medyczne Oporow, Wroclaw, Lower Silesian Voivodeship
  - OKOLEK, Wroclaw, Lower Silesian Voivodeship
  - EuroMediCare Szpital Specjalistyczny z Przychodnia we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - lnstytut Gruzlicy i Chorob Pluc, Warsaw, Masovian Voivodeship
  - Spoldzielnia Pracy Lekarzy Specjalistow Medicus (for OCT), Szczecin, West Pomeranian Voivodeship
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Przychodnia EVOMED Pracownia USG i RTG, Szczecin, West Pomeranian Voivodeship
  - Centrum Pulmonologii i Torakochirurgii w Bystrej (DLCO), Bystra
  - Centrum Medyczne Ksiezy Mlyn sp. z o.o. (Ophtalmoscopy, OCT), Lodz
  - Centra Medyczne 'MEDYCEUSZ" (Chest X-Ray), Lodz
  - Wojewodzki Szpital Specjalistyczny im.dr. WI. Bieganskiego (endoscopy), Lodz
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - MEDICOME- Oswiecimskie Centrum Medyczne (OCT), Oświęcim
  - Centrum Zdrowia MDM, Warsaw
  - Endomed, Wroclaw
  - Amicare Sp. z o.o. Sp.k., Lodz, Łódź Voivodeship
  - IP Clinic Sp. z o.o., Lodz, Łódź Voivodeship
- Centro Hospitalar Universitario de Sao Joao, E.P.E, Porto, Portugal
- Russia (18):
  - "Clinic Ultrasound 4D" LLC, Pyatigorsk, Stavropol Kray
  - "Platnaya poliklinika" LLC, Pyatigorsk, Stavropol Kray
  - SBHI of Nizhniy Novgorod region "Nizhniy Novgorod Regional Clinical Hospital n.a. N.A. Semashko, Nizhny Novgorod
  - BHI of Omsk region "Clinical oncology dispensary", Omsk
  - Clinicodiagnostic center "Ultramed", Omsk
  - Medical center "Intervzglyad", Omsk
  - FSBEI of Higher Education "North-Western State Medical University n.a. I.I. Mechnikov" of MoH RF, Saint Petersburg
  - FSBEI of Higher Education "I.P.Pavlov First Saint Petersburg State Medical University" of MoH of RF, Saint Petersburg
  - Private Institution, Educational Organization of Higher Education "Medical University "Reaviz", Samara
  - Private Institution, Educational Organization of Higher Education "Medical University "Reaviz",, Samara
  - Clinical Hospital Russian Railways - Medicina, Samara
  - Medical Company "Hepatolog" LLC, Samara
  - Samara Diagnostic center, Samara
  - Regional Medical center LLC (Branchevsky's clinic), Samara
  - Inter-branch scientific and technical complex "Eye microsurgery", Smolensk
  - Multidisciplinary Medical center "Clinic Park", Smolensk
  - "Uromed" LLC, Smolensk
  - Autonomous Noncommercial Medical Organization "Stavropol Regional Clinical Advisory-Diagnostic, Stavropol
- South Korea (11):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Endoscopy Facility in kyungpook National University Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - OCT Facility In kyungpook Natioanl University Hospital, Daegu
  - PFT Facility in kyungpook Natioanl University Hospital, Daegu
  - Endoscopy Facility in Severance Hospital, Yonsei University Health System, Seoul
  - OCT(1) Facility in Severance Hospital, Yonsei University Health System, Seoul
  - OCT(2) Facility in Severance Hospital, Yonsei University Health System, Seoul
  - PFT(1) Facility Severance Hospital, Yonsei University Health System, Seoul
  - PFT(2) Facility Severance Hospital, Yonsei University Health System, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Hospital Universitario la Paz, Madrid, Spain
- Ukraine (17):
  - Limited Liability Company "Lookout "Medical Center", Dnipro
  - Limited Liability Company "MDC EXPERT", Dnipro
  - Municipal Enterprise <<Dnipro Reg Clinical Hosp named after M. I.I. Mechnikov>>, Dnipro
  - Clinical Diagnostical Center "Simedgroup", Ivano-Frankivsk
  - CNE Regional Clinical Hospital of Ivano-Frankivsk Regional Council,Department of Gastroenterology, Ivano-Frankivsk
  - Llc "Ldts-Skaymed", Kharkiv
  - CNE Prof. O.O. Shalimov City Clinical Hospital #2 of Kharkiv City Council, Department of Proctology, Kharkiv
  - Llc Medical Center Oftalmika, Kharkiv
  - CNE Kyiv City Clinical Hospital #1 of Executive Body of Kyiv City Council (Kyiv City State, Kyiv
  - Transcarpathian Center of Eye Microsurgery, Uzhhorod
  - CNE Andrii Novak Transcarpathian Regional Clinical Hospital of, Uzhhorod
  - Medical Center of LLC Health Clinic, Med Clinical lnvestigational Center, Unit of Gastroenterology,, Vinnytsia
  - CNE "Vinnytsia Reg Clinical Hosp named after N.I.Pirogov Vinnytsia Regional Council", Reg Specialize, Vinnytsia
  - Podilskyi tsentr zoru, Vinnytsia
  - Scientific and Research Institute of lnvalid Rehabilitation (Educational and Scientific, Vinnytsia
  - Diagnostic Center "Mediscan", Vinnytsia
  - Llc "Optimal M", Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD334-210

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 234 participants with moderately active ulcerative colitis (UC) were enrolled in the study.
Groups:
- Etrasimod: Participants with moderately active UC were randomized to receive Etrasimod 2 milligrams (mg) tablet orally once daily (QD) for 52-Week.
- Placebo: Participants with moderately active UC were randomized to receive placebo matched to Etrasimod tablet orally QD for 52-Week.
Period: Overall Study
Arm/Group | Etrasimod | Placebo
Started | 155 | 79
Safety Set | 154 | 79
Primary Analysis Set | 127 | 60
Completed | 97 | 34
Not Completed | 58 | 45
Not completed — Adverse Event | 8 | 2
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Physician Decision | 2 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Participant terminated by sponsor | 1 | 0
Not completed — Disease worsening | 36 | 36
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Etrasimod: Participants with moderately active UC were randomized to receive Etrasimod 2 mg tablet orally QD for 52-Week.
- Total: Total of all reporting groups
Arm/Group | Etrasimod | Placebo | Total
Number analyzed (Participants) | 154 | 79 | 233
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (13.15) | 40.8 (13.00) | 41.3 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 40 | 103
  Male | 91 | 39 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 146 | 73 | 219
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 143 | 67 | 210
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Remission (CR) at Week 52 Using Modified Mayo Score (MMS)
Description: MMS is used to assess disease activity in participants with UC and has following components: endoscopic score(ES),rectal bleeding(RB),stool frequency(SF).Each component score ranges from 0 to 3(0=normal,1=mild,2=moderate,3=severe); higher scores indicating more severe disease.ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy,scores ranged from 0(normal or inactive disease) to 3(severe disease [spontaneous bleeding, ulceration]).RB reported most severe amount of blood passed per rectum in 24-hour period,scores ranged from 0(no blood seen) to 3(blood alone passes).SF reported number of stools in 24-hour period relative to normal number of stools for that participant in same period,scores ranged from 0(normal number of stools) to 3(5 or more stools than normal).CR per FDA draft guidance defined as:SF=0 or 1 and no greater than baseline, RB=0,ES less than or equal to (<=)1(excluding friability).Percentage of participants achieving CR at Week 52 was evaluated.
Time Frame: Week 52
Population: Primary analysis set included all randomized participants who received at least 1 dose of study treatment with baseline MMS [total score range: 0 to 9, higher score = more severity] 4-6, baseline ES greater than or equal to (>=2) and baseline RB score >=1.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 26.0 | 18.3
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; Difference (%) for etrasimod minus placebo was based on estimated common risk difference using the Mantel- Haenszel weights. The 2-sided p-value was used to test the hypothesis of the risk difference being 0; Test type: Superiority; p = 0.2524, Mantel Haenszel; Risk Difference (RD) = 7.35, 95% CI 2-sided [-5.24 to 19.94]

2. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Week 12 Using MMS
Description: MMS is used to assess disease activity in participants with UC and has following components: ES, RB and SF. Each component score ranges from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe); higher scores indicating more severe disease. ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, scores ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]). RB reported the most severe amount of blood passed per rectum in a 24-hour period, scores ranged from 0 (no blood seen) to 3 (blood alone passes). SF reported number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, score ranged from 0 (normal number of stools) to 3 (5 or more stools than normal). CR per FDA draft guidance was defined as: SF=0 or =1 and no greater than baseline, RB=0, and ES <=1 (excluding friability). Percentage of participants achieving CR at Week 12 was evaluated in this endpoint.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 28.3 | 11.7
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; Difference (%) for etrasimod minus placebo was based on estimated common RD using the Mantel- Haenszel weights. The 2-sided p-value was used to test the hypothesis of the RD being 0; Test type: Superiority; p = 0.0068, Mantel Haenszel; Risk Difference (RD) = 15.61, 95% CI 2-sided [4.31 to 26.91]

3. Secondary Outcome: Percentage of Participants Achieving Endoscopic Improvement at Week 52
Description: Endoscopic improvement was defined as ES <=1 (excluding friability). ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]), higher scores = more severity. Percentage of participants achieving endoscopic improvement at Week 52 was evaluated in this endpoint.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 32.3 | 23.3
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2302, Mantel Haenszel; Risk Difference (RD) = 8.24, 95% CI 2-sided [-5.22 to 21.71]

4. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission at Week 52
Description: Symptomatic remission was defined as SF =0 (or = 1 with a >= 1 point decrease from baseline) and RB =0. SF subscore: reported number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, scores ranged from 0 (normal number of stools) to 3 (5 or more stools than normal), higher scores = more severity. RB subscore: reported the most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0 (no blood seen) to 3 (blood alone passes), higher scores = more severity. Percentage of participants achieving symptomatic remission at Week 52 was evaluated in this endpoint.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 37.0 | 30.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; Difference (%) for etrasimod minus placebo was based on estimated common RD using the Mantel- Haenszel weights, where only participants with an assessment at Baseline and the corresponding visit are included. The 2-sided Nominal p-value was used to test the hypothesis of the RD being 0; Test type: Superiority; p = 0.3339, Mantel Haenszel; Risk Difference (RD) = 7.12, 95% CI 2-sided [-7.32 to 21.55]

5. Secondary Outcome: Percentage of Participants Achieving Complete Symptomatic Remission at Week 52
Description: Complete symptomatic remission was defined as participants with RB = 0 and SF = 0. SF subscore: reported number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, scores ranged from 0 (normal number of stools) to 3 (5 or more stools than normal), higher scores = more severity. RB subscore: reported the most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0 (no blood seen) to 3 (blood alone passes), higher scores = more severity. Percentage of participants achieving complete symptomatic remission at Week 52 was evaluated in this endpoint.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 20.5 | 20.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.9141, Mantel Haenszel; Risk Difference (RD) = 0.68, 95% CI 2-sided [-11.76 to 13.13]

6. Secondary Outcome: Percentage of Participants Achieving Histologic-Endoscopic Mucosal Improvement at Week 52
Description: Histologic-endoscopic mucosal improvement was defined as ES <=1 (excluding friability) with Geboes score <2.0. ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]), higher scores = more severity. The Geboes score grading system was a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicated more severe disease. Percentage of participants achieving mucosal improvement at Week 52 was evaluated in this endpoint.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 25.2 | 15.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1089, Mantel Haenszel; Risk Difference (RD) = 9.56, 95% CI 2-sided [-2.13 to 21.25]

7. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Both Weeks 12 and 52 [Combined] Using MMS
Description: MMS is used to assess disease activity in participants with UC and has following components: ES, RB and SF. Each component score ranges from 0 to 3 (0= normal, 1= mild, 2= moderate, 3= severe); higher scores = more severe disease. ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0 (normal or inactive disease) to 3 (severe disease). RB: reported the most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0 (no blood seen) to 3 (blood alone passes). SF reported number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, score ranged from 0 (normal number of stools) to 3 (5 or more stools than normal). Clinical remission per FDA draft guidance: SF =0 or =1 and no greater than baseline, RB =0, and ES <=1 (excluding friability). Percentage of participants who achieved clinical remission at both the time points Week 12 and Week 52 [Combined] are reported.
Time Frame: Weeks 12 and 52 [Combined]
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 16.5 | 5.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0104, Mantel Haenszel; Risk Difference (RD) = 11.19, 95% CI 2-sided [2.63 to 19.75]

8. Secondary Outcome: Percentage of Participants With 12-Week Corticosteroid-Free Clinical Remission at Week 52 Among Participants Receiving Corticosteroids at Baseline Using MMS
Description: MMS has following components:ES, RB and SF. Each component score ranges from 0 to 3(0=normal,1=mild,2=moderate,3=severe); higher scores indicating more severe disease. ES:worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0(normal or inactive disease)to 3(severe disease). RB:most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0(no blood seen)to 3(blood alone passes). SF:number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, score ranged from 0(normal number of stools)to 3(5 or more stools than normal). CR per FDA draft guidance as: SF =0 or =1 and no greater than baseline, RB=0, and ES <=1(excluding friability). 12-week corticosteroid-free CR was defined as CR at Week 52 and corticosteroid-free for >=12 weeks immediately prior to Week 52. The baseline was balanced between treatment groups and representative of participants with mildly to moderately active UC.
Time Frame: Week 52
Population: Primary analysis set included all randomized participants who received at least 1 dose of study treatment with baseline MMS [total score range: 0 to 9, higher score = more severity] 4-6, baseline ES greater than or equal to (>=2) and baseline RB score >=1. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who received oral corticosteroids for UC at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 37 | 18
Percentage of participants | 16.2 | 16.7
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9203, Mantel Haenszel; Risk Difference (RD) = -1.07, 95% CI 2-sided [-22.06 to 19.92]

9. Secondary Outcome: Percentage of Participants With 12-Week Corticosteroid-Free Clinical Remission at Week 52 Using MMS
Description: MMS has following components: ES, RB and SF. Each component score ranges from 0 to 3 (0=normal,1=mild,2=moderate,3=severe); higher scores indicating more severe disease. ES: worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0(normal or inactive disease) to 3 (severe disease). RB: most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0(no blood seen) to 3 (blood alone passes). SF: number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, score ranged from 0(normal number of stools) to 3 (5 or more stools than normal). CR per FDA draft guidance as: SF =0 or =1 and no greater than baseline, RB=0, and ES <=1(excluding friability). 12-week corticosteroid-free CR was defined as CR at Week 52 and corticosteroid-free for >=12 weeks immediately prior to Week 52.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 25.2 | 16.7
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1726, Mantel Haenszel; Risk Difference (RD) = 8.49, 95% CI 2-sided [-3.71 to 20.68]

10. Secondary Outcome: Percentage of Participants Achieving 4-Week Corticosteroid-Free Clinical Remission at Week 52 Among Participants Receiving Corticosteroids at Baseline Using MMS
Description: MMS has following components: ES, RB and SF; each ranged as 0=normal,1=mild,2=moderate,3=severe; total MMS score 0-9; higher scores=more severe disease. ES:worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0(normal or inactive disease)to 3(severe disease). RB:most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0(no blood seen) to 3(blood alone passes). SF:number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, score ranged from 0(normal number of stools)to 3(5 or more stools than normal). CR per FDA draft guidance as: SF =0 or =1 and no greater than baseline, RB=0, and ES <=1(excluding friability). 4-week corticosteroid-free CR was defined as CR at Week 52 and corticosteroid-free for >=4 weeks immediately prior to Week 52. The baseline was balanced between treatment groups and representative of participants with mildly to moderately active UC.
Time Frame: Week 52
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 20 | 10
Percentage of participants | 30.0 | 30.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9272, Mantel Haenszel; Risk Difference (RD) = -1.71, 95% CI 2-sided [-38.31 to 34.90]

11. Secondary Outcome: Percentage of Participants With 4-Week Corticosteroid-Free Clinical Remission at Week 52 Using MMS
Description: MMS has following components: ES, RB and SF. Each component score ranges from 0 to 3 (0=normal,1=mild,2=moderate,3=severe); where total score is sum of three components giving total MMS score as 0 to 9; higher scores indicating more severe disease. ES: worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0(normal or inactive disease) to 3 (severe disease). RB: most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0(no blood seen) to 3 (blood alone passes). SF: number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, score ranged from 0 (normal number of stools) to 3 (5 or more stools than normal). CR per FDA draft guidance as: SF =0 or =1 and no greater than baseline, RB=0, and ES <=1(excluding friability). 4-week corticosteroid-free CR was defined as CR at Week 52 and corticosteroid-free for >=4 weeks immediately prior to Week 52.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 25.2 | 16.7
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1726, Mantel Haenszel; Risk Difference (RD) = 8.49, 95% CI 2-sided [-3.71 to 20.68]

12. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 12 Using MMS
Description: Clinical response was defined as a >=2-point and >=30 percentage (%) decrease from baseline in MMS, and a >=1-point decrease from baseline in RB subscore or an absolute RB subscore <=1 and is as per FDA draft guidance. MMS was used to assess disease activity in participants with UC and has following components: ES, RB and SF. Each component score ranges from 0 to 3 (0= normal, 1= mild, 2= moderate, 3= severe); where total score is sum of three components giving total MMS score as 0 to 9; higher scores indicating more severe disease. ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]). Percentage of participants achieving clinical response at Week 12 was evaluated in this endpoint.
Time Frame: Week 12
Population: Primary analysis set included all randomized participants who received at least 1 dose of study treatment with baseline MMS 4-6, baseline ES >=2 and baseline RB score >=1.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 55.9 | 36.7
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0151, Mantel Haenszel; Risk Difference (RD) = 18.64, 95% CI 2-sided [3.61 to 33.67]

13. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 52 Using MMS
Description: Clinical response was defined as a >=2-point and >=30 % decrease from baseline in MMS, and a >=1-point decrease from baseline in RB subscore or an absolute RB subscore <=1 and is as per FDA draft guidance. MMS is used to assess disease activity in participants with UC and has following components: ES, RB and SF. Each component scores ranges from 0 to 3 (0= normal, 1= mild, 2= moderate, 3= severe); where total score is sum of three components giving total MMS score as 0 to 9; higher scores indicating more severe disease. ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, scores ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]). Percentage of participants achieving clinical response at Week 52 was evaluated in this endpoint.
Time Frame: Week 52
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 44.1 | 38.3
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4419, Mantel Haenszel; Risk Difference (RD) = 5.96, 95% CI 2-sided [-9.22 to 21.13]

14. Secondary Outcome: Percentage of Participants Achieving Endoscopic Improvement at Week 12
Description: Endoscopic improvement was defined as ES <=1 (excluding friability). ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, scores ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]), higher scores = more severity. Percentage of participants achieving endoscopic improvement at Week 12 was evaluated in this endpoint.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 44.1 | 20.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0007, Mantel Haenszel; Risk Difference (RD) = 23.33, 95% CI 2-sided [9.78 to 36.89]

15. Secondary Outcome: Percentage of Participants Achieving Histologic-Endoscopic Mucosal Improvement at Week 12
Description: Histologic-endoscopic mucosal improvement was defined as ES <=1 (excluding friability) with Geboes score <2.0. ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, scores ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]), higher scores = more severity. The Geboes score grading system was a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicated more severe disease. Percentage of participants achieving mucosal improvement at Week 12 was evaluated in this endpoint.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 29.1 | 13.3
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0128, Mantel Haenszel; Risk Difference (RD) = 14.99, 95% CI 2-sided [3.19 to 26.79]

16. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission at Week 12
Description: Symptomatic remission was defined as SF =0 (or = 1 with a >= 1 point decrease from baseline) and RB =0. SF subscore: reported number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, scores ranged from 0 (normal number of stools) to 3 (5 or more stools than normal), higher scores = more severity. RB subscore: reported the most severe amount of blood passed per rectum in a 24-hour period, scores ranged from 0 (no blood seen) to 3 (blood alone passes), higher scores = more severity. Percentage of participants achieving symptomatic remission at Week 12 was evaluated in this endpoint.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 36.2 | 25.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1492, Mantel Haenszel; Risk Difference (RD) = 10.24, 95% CI 2-sided [-3.67 to 24.14]

17. Secondary Outcome: Percentage of Participants Achieving Complete Symptomatic Remission at Week 12
Description: Complete symptomatic remission was defined as participants with RB = 0 and SF = 0. SF subscore: reported number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, scores ranged from 0 (normal number of stools) to 3 (5 or more stools than normal), higher scores = more severity. RB subscore: reported the most severe amount of blood passed per rectum in a 24-hour period, scores ranged from 0 (no blood seen) to 3 (blood alone passes), higher scores = more severity. Percentage of participants achieving complete symptomatic remission at Week 12 was evaluated in this endpoint.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 20.5 | 20.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.9774, Mantel Haenszel; Risk Difference (RD) = 0.18, 95% CI 2-sided [-12.18 to 12.53]

18. Secondary Outcome: Percentage of Participants Achieving Change From Baseline in Both ES and RB or in Both ES and SF at Week 12
Description: ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, scores ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]), higher scores = more severity. RB: reported the most severe amount of blood passed per rectum in a 24-hour period, scores ranged from 0 (no blood seen) to 3 (blood alone passes), higher scores = more severity. SF reported number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, score ranged from 0 (normal number of stools) to 3 (5 or more stools than normal), higher scores = more severity. Percentage of participants with reduction from baseline in both ES and RB or in both ES and SF at Week 12 was evaluated in this endpoint. The baseline primary analysis set was balanced between treatment groups and representative of participants with mildly to moderately active UC.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 44.9 | 21.7
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0011, Mantel Haenszel; Risk Difference (RD) = 22.83, 95% CI 2-sided [9.17 to 36.49]

19. Secondary Outcome: Percentage of Participants Achieving Histologic Response Based on the Geboes Grading System at Week 12
Description: Histologic response based on the Geboes grading system was defined as Geboes score <=3.1. The Geboes score grading system is a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicated more severe disease. Percentage of participants achieving histologic response based on the Geboes grading system at week 12 was evaluated in this endpoint.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 44.9 | 33.3
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1513, Mantel Haenszel; Risk Difference (RD) = 10.8, 95% CI 2-sided [-3.95 to 25.56]

20. Secondary Outcome: Percentage of Participants Achieving Histologic Response Based on Robarts Histopathology Index (RHI) at Week 12
Description: RHI is an evaluative index, derived from the Geboes score, that is designed to be reproducible and responsive to clinically meaningful change in disease activity over time. Histologic response based on RHI was defined as decrease in RHI of >=7 points from baseline. Total RHI score ranges from 0 (no disease activity) to 33 (severe disease activity), higher score = more severity. Percentage of participants achieving histologic response based on RHI at Week 12 was evaluated in this endpoint.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 127 | 60
Percentage of participants | 46.5 | 35.0
Statistical Analysis 1: Comparison: Etrasimod vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1823, Mantel Haenszel; Risk Difference (RD) = 10.07, 95% CI 2-sided [-4.73 to 24.87]

21. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and all non-SAEs.
Time Frame: From first dose of study treatment up to 4 weeks post last dose of study treatment (up to 56 Weeks)
Population: Safety set included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 154 | 79
Participants | 101 | 49

22. Other Pre Specified Outcome: Number of Participants With AEs Based on Severity
Description: An AE was any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Severity was classified using common terminology criteria for adverse events (CTCAE), version 5.0, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death related to AE. Only those categories in which at least 1 participant had data for any reporting group were reported.
Time Frame: From first dose of study treatment up to 4 weeks post last dose of study treatment (up to 56 Weeks)
Population: Safety set included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrasimod | Placebo
Number analyzed (Participants) | 154 | 79
Participants
  Grade 1 | 48 | 23
  Grade 2 | 42 | 24
  Grade 3 | 11 | 2

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 4 weeks post last dose of study treatment (up to 56 Weeks)
Description: Same event may occur as both non-SAE and SAE but are distinct events. An event may be categorised as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety set included all randomised participants who received at least 1 dose of study treatment.
Arm/Group | Etrasimod | Placebo
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/79
Serious Adverse Events (participants affected / at risk) | 10/154 | 1/79
Other Adverse Events (participants affected / at risk) | 100/154 | 48/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etrasimod (N=154) | Placebo (N=79)
Colitis ulcerative (Gastrointestinal disorders) | 4 (4) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etrasimod (N=154) | Placebo (N=79)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 6 (6)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Splenic cyst (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (2) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Epiretinal membrane (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid thickening (Eye disorders) | 1 (1) | 0 (0)
Floppy eyelid syndrome (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (2) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 19 (19) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophageal polyp (Gastrointestinal disorders) | 0 (0) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1)
Early satiety (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 5 (5) | 0 (0)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 3 (4) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 15 (16) | 7 (7)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 3 (3)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (15) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (10) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (4) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1)
Blood cholesterol increased (Investigations) | 3 (4) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 5 (5) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 2 (2) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (2) | 0 (0)
Blood triglycerides increased (Investigations) | 8 (9) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 1 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 13 (20) | 2 (2)
Heart rate decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0)
Lung diffusion test decreased (Investigations) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (5) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 2 (2)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (7) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 3 (3)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Crystalluria (Renal and urinary disorders) | 1 (1) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 2 (4) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Skin fibrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Postmenopause (Social circumstances) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT04607837/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04607837/SAP_001.pdf